CLINICAL TRIAL: NCT00398632
Title: Switching to Duloxetine to Ameliorate SSRI-Induced Sexual Dysfunction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit subjects
Sponsor: Stanford University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Lorrin M Koran, Professor of Psychiatry, Emeritus, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 97143
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Results first posted 2015-06-16 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine (Experimental): Duloxetine 60 mg, by mouth, once daily or twice daily (as needed to control symptoms of major depression)
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — dosage form: capsule. dosage: 60 mg. frequency: once daily, or twice daily if 120 mg/day is needed to control symptoms of major depression. duration: 12 weeks
  Other Names: Cymbalta

SUMMARY:
Sexual dysfunction is a common side effect of selective serotonin reuptake inhibitors (SSRIs). The hypotheses of this study are that:1. subjects with major depression or dysthymia who are being treated with an SSRI and experiencing treatment-related sexual dysfunction will experience less sexual dysfunction if they are switched to duloxetine, and 2. they will experience either improved antidepressant response or no loss of antidepressant response.

DETAILED DESCRIPTION:
In this study, subjects suffering from depression or dysthymia and experiencing treatment-emergent sexual dysfunction from an SSRI are switched from their SSRI to duloxetine to determine whether or not they experience improved sexual function and equal or improved antidepressant response. Study subjects are assigned to receive open label duloxetine for 12 weeks at either 60mg per day or 120mg per day after discontinuing their current antidepressant

ELIGIBILITY:
Inclusion Criteria::

* age 18 - 65 inclusive
* able to read and understand informed consent
* informed consent given
* currently being treated with an SSRI for depression or dysthymia
* currently suffering from treatment-emergent sexual dysfunction attributable to the SSRI
* have normal safety lab values at screen
* if currently taking medication to improve sexual performance, willing to discontinue the drug for the duration of the study
* female subjects of child bearing age need to use an acceptable form of birth control throughout the study Exclusion Criteria:- being pregnant, breastfeeding, or planning to become pregnant within 4 months
* suffering from psychotic, substance abuse, bipolar, or organic mental disorder, OCD, panic disorder, or personality disorder severe enough to interfere with study participation
* suffer from an unstable or serious medical disorder
* having a medical disorder that could be the cause of the sexual dysfunction
* taking a medication that is metabolized by hepatic enzyme CYP2D6
* having used a MAOI within 15 days of proposed start of duloxetine treatment
* having a known hypersensitivity to duloxetine or any of its ingredients
* having taken viagra or related drug within 3 months prior to starting SSRI treatment
* requiring ongoing treatment with a mood stabilizer (anticonvulsant) or antipsychotic medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-11; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorrin M Koran, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine
Started | 6
Completed | 4 (2/6 subjects withdrew at end of week 6; 1 for lack of efficacy, 1 because of time constraints.)
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Population: Adult patients taking an antidepressant drug and troubled by sexual side effects of the drug
Groups:
- Duloxetine: Duloxetine: dosage form: capsule. dosage: 60 mg. frequency: once daily, or twice daily if 120 mg/day is needed to control symptoms of major depression. study duration: 12 weeks
Arm/Group | Duloxetine
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean age only. The data were destroyed some years ago, and only the mean age was preserved.
  years | 44 (NA) — The data were destroyed some years ago, and only the mean age was preserved.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 6
Antidepressant taken prior to duloxetine switch [Number; unit: participants]
  venlafaxine | 3
  citalopram | 2
  fluoxetine | 1
Clinically Depressed [Count of Participants; unit: Participants] — Patients with score >22 assessed by Inventory for Depressive Symptomology-Clinician Rated (IDS-C). The IDS-C is a 30-item inventory designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes.
  Participants | 2

OUTCOME MEASURES:

1. Primary Outcome: Global Clinical Impressions Improvement Score re Sexual Functioning
Description: The GCI-I score is a global clinical impression score regarding a patient's symptom severity change rated by the treating clinician. The score can be 0 (not assessed), 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse) or 7 (very much worse). In this study clinicians made ratings based on interviewing the patient and reviewing the patient's self ratings on the the Arizona Sexual Experiences Scale (ASEX). No formal cut point scores on the ASEX were established. The ASEX is a 5-item slef rating scale that quantifies sex drive, arousal, vaginal lubrication/penile erection, ability to reach organism, and satisfaction from orgasm. Each item is rated from 1 to 6 (total scores from 5 to 30), with higher scores indicating greater sexual dysfunction.
Time Frame: baseline and last observation (4 subjects at end of week 12, 2 subjects at end of week 6)
Population: Four subjects completed the study; two withdrew at end of week six. CGI-I ratings for two subjects were done at end of week 6 and this last observation was carried forward in the analysis. CGI-I ratings for the 4 completing subjects were done at end of week 12.
Measure: Number; unit: participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 6
participants
  CGI sexual functioning much improved | 1
  CGI sexual functioning minimally improved | 3
  CGi-I sexual functioning unchanged | 1
  CGI sexual functioning much worse | 1

2. Secondary Outcome: Count of Patients With Remission of Depressive Symptoms According to the Inventory for Depressive Symptomology-Clinician Rated (IDS-C) at End of Study
Description: The IDS-C is a 30-item inventory designed to assess the severity of depressive symptoms. Scale range minimum = 0 / maximum = 84. Higher values are considered to be worse outcomes. Scores less than or equal to 6 indicated remission in this study.
Time Frame: Last observation (4 subjects at end of week 12, 2 subjects at end of week 6)
Population: All participants; the last observed non-missing value was used (LOCF)
Measure: Count of Participants; unit: Participants
Arm/Group | Duloxetine
Number analyzed (Participants) | 6
Participants | 5

ADVERSE EVENTS:
Arm/Group | Duloxetine
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Open label trial, only six subjects enrolled, only 4 completed the trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No